CLINICAL TRIAL: NCT05649423
Title: Effects of Postural Drainage With and Without Percussion on Mucus Clearance, Dyspnea and Quality of Life in Chronic Obstructive Pulmonary Disease
Brief Title: Postural Drainage With and Without Percussion in Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/ 0349 Zunaira Zaheer
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, Mucus, Dyspnea, cough, postural drainage, percussion
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Cough | interventions — Drainage, Postural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postural drainage with percussion (Experimental): Chest percussion is performed with cupped hands in an alternating rhythmic manner The force applied must be equal 8 weeks, 3 sessions per week , each session took about 30 minutes
  Interventions: Other: POSTURAL DRAINAGE WITH PERCUSSION; Other: Postural drainage
- Postural drainage (Active Comparator): Postural drainage without Percussion Each position should be held for a minimum of five minutes Use pillows, foam wedges for comfort make position on patient back, side and stomach 8 weeks, 3 sessions of alternating positions per , each session took about 30 minutes
  Interventions: Other: Postural drainage

INTERVENTIONS:
Other: POSTURAL DRAINAGE WITH PERCUSSION — Each position should be held for a minimum of five minutes. In each position, your chest should be lower than your hips to allow mucus to drain. On your back: Patient's chest should be lower than his hips, which you can achieve by lying on a slanted surface up about 18 to 20 inches. On your sides: With pillows under your hips, lie on one side. To clear congestion from the right and left lobes. On your stomach: Drape patient's body over a stack of pillows, this is best in clearance of mucus from the lower back area of the lungs.
  Percussion The equipment required here is cupped hands of caregiver to deliver the force required to drain the thick secretions. Patient should be in a comfortable position to enhance the effect. This loosens the thick, sticky secretions from the walls of the lung allowing them to into the larger airways, The sound heard must be hollow. The force applied must be equal.
  Arms: Postural drainage with percussion
Other: Postural drainage — * Each position should be held for a minimum of five minutes.
  * In each position, your chest should be lower than your hips to allow mucus to drain On your back: Patient's chest should be lower than your hips, which you can achieve by lying on a slanted surface or propping patient's hips up about 18 to 20 inches
  * This position is best for draining the bottom front parts of your lungs. On your sides: With pillows under your hips, lie on one side so that your chest is lower than your hips. To clear congestion from the bottom part of the right lung, lie on your left side. To clear congestion from the bottom part of your left lung, lie on your right side.
  On your stomach: Drape patient's body over a stack of pillows or other object, and rest his arms by his head, with his chest lower than his hips. This position is best for clearing mucus in the lower back area of the lungs.

SUMMARY:
Effects Of postural drainage with and without percussion on mucus clearance, dyspnea and quality of life in Chronic Obstructive Pulmonary disease. 34 Patients will be explained in detail about the procedure under study. Informed consent will be taken.

Subjects will be evaluated using the Modified medical research council and Dyspnea-12 Questionnaire for (dyspneal), St George's Respiratory Questionnaire for quality of life. Cough and Sputum assesment questionnaire for mucus clearance would be used. One group will be tested by Postural drainage techniques and the second group will be tested by Postural drainage with Percussion.

DETAILED DESCRIPTION:
Chronic respiratory diseases refer to chronic diseases of the airways and other structures like alveoli bronchi and bronchioles of the lung. Some of the most common diseases include asthma, chronic obstructive pulmonary disease (COPD), and other respiratory allergies. COPD leads to permanent damaged airways, which causes them to become narrower making it difficult for air to go into and out of lungs it belongs to a group of progressive lung diseases that make it difficult to breathe - including chronic bronchitis and emphysema (assessed by pulmonary function and x-ray evidence).

People have difficulty breathing due to long-term damage to their lungs, caused mainly due to cigarette smoking, exposure to air pollution, exposure to fumes or particles at work, for example, welding fumes or coal dust and Alpha-1-antitrypsin deficiency, a genetic condition. Symptoms that badly effects the health of the patient includes cough, decreased exercise tolerance production, shortness of breath, and shortness of breath.

In this research, the effects of postural drainage with and without percussion on mucus clearance, dyspnea and quality of life would be determined. Chest physiotherapy is the term for a group of treatments designed to eliminate secretions, thus helping to decrease work of breathing, promote the expansion of the lungs, and prevent the lungs from collapse.

There is a large impact on quality of life for individuals living with COPD, decreased exercise tolerance, decreased ability to carry out activities of daily living (ADLs), anxiety, feelings of isolation, decreased social participation etc.

This study will be a randomized controlled trial. The study will be conducted in Sheikh Zaid hospital Lahore. In the present study under considerations we mainly look on the subjects meeting predetermined inclusion and exclusion criteria will be divided into two groups using lottery method. Sample size will be 34 which would include both male and female. Subjects irrespective of gender aged between 35-65 years of age are involved.

ELIGIBILITY:
Inclusion Criteria:

* • Age 35-65 years

  * Patients who have had exacerbations in the past month
  * Agreeing to participate in the study after having provided a written consent.
  * Patients with heavy Mucus secretions in Lungs Field
  * Diagnosed Patients of Chronic Obstructive Pulmonary Disease Stage 2(COPD)

Exclusion Criteria:

* • Patients on bronchodilators and steroids

  * Patients with severe Pulmonary Edema
  * Patients with severe rib fractures
  * History of any recent thoraco abdominal surgery(35)
  * Left ventricular Ejection Fraction (EF)
  * Anemic patients
  * Pregnant women

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
For Airway Clearance | 8weeks
  Sputum diary Questionnaire will be used
St. George's Respiratory Questionnaire (SGRQ) quality of life assessment | 8 weeks
  For assessment and changes in Quality of life Questionnaire will be used
Spirometry For Airway clearance | 8 weeks
  Spirometer will be used for evaluating the Forced Expiratory values in 1 second

OTHER OUTCOMES:
Dyspnea-12 | 8 weeks
  Dyspnea-12 questionnaire is used to check for the dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Sumera Abdulhameed, MS, Principal Investigator — Riphah International University
Locations (1):
- Sheikh Zaid Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No